CLINICAL TRIAL: NCT03215524
Title: A Randomized Phase II, Open Label, Study of Daratumumab, Weekly Low-Dose Oral Dexamethasone and Cyclophosphamide With or Without Pomalidomide in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study Of Daratumumab, Low-Dose Oral Dexamethasone and Cyclophosphamide With Or Without Pomalidomide
Acronym: DCDP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Myeloma Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMRG 004
Record Dates: First submitted 2017-06-05; First posted 2017-07-12 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — 2'-deoxycytidine diphosphate; daratumumab; Cyclophosphamide; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (Experimental): Daratumumab, Cyclophosphamide, Dexamethasone, Pomalidomide
  Daratumumab, IV, at 16 mg/kg, or Daratumumab, SC, at 1800 mg on days 1, 8, 15 and 22 for Cycles 1 and 2, on Days 1 and 15 for Cycles 3-6, and Day 1 of each cycle for Cycle 7 and beyond for each 28-day cycle.
  Cyclophosphamide, orally, at 400 mg on Days 1, 8, 15 of each 28-day cycle for 24 cycles.
  Dexamethasone, orally, at 20 mg on day of daratumumab administration (pre-daratumumab) and 20 mg on the following day. On weeks without daratumumab administration, 40 mg dexamethasone weekly.
  Pomalidomide, orally, at 4 mg on Days 1- 21 of each 28-day cycle.
  Interventions: Biological: DCdP
- ARM B (Experimental): Daratumumab, Cyclophosphamide, Dexamethasone, Pomalidomide
  Daratumumab, IV, at 16 mg/kg, or Daratumumab, SC, at 1800 mg on days 1, 8, 15 and 22 for Cycles 1 and 2, on Days 1 and 15 for Cycles 3-6, and Day 1 of each cycle for Cycle 7 and beyond for each 28-day cycle.
  Cyclophosphamide, orally, at 400 mg on Days 1, 8 and 15 of each 28-day cycle for 24 cycles.
  Dexamethasone,orally, at 20 mg on day of daratumumab administration (pre-daratumumab) and 20 mg on the following day. On weeks without daratumumab administration,40mg dexamethasone weekly.
  Pomalidomide, orally, added at first progression at 4 mg on Days 1- 21 of each 28-day cycle.
  Interventions: Biological: DCd+P

INTERVENTIONS:
Biological: DCdP — Daratumumab, Cyclophosphamide, Dexamethasone, Pomalidomide
  Other Names: Darzalex; Cytoxan; Pomalyst; Daratumumab; Cyclophosphamide; Pomalidomide; Dexamethasone
  Arms: ARM A
Biological: DCd+P — Daratumumab, Cyclophosphamide, Dexamethasone, + Pomalidomide added only at first confirmed biochemical progression
  Other Names: Darzalex; Cytoxan; Pomalyst; Daratumumab; Cyclophosphamide; Dexamethasone
  Arms: ARM B

SUMMARY:
This is a randomized phase II open label study of daratumumab, weekly low-dose oral cyclophosphamide and dexamethasone with or without pomalidomide in patients with relapsed and refractory multiple myeloma. The study consists of two arms. Patients will be randomized into ARM A and ARM B in a 1:1 ratio.

DETAILED DESCRIPTION:
This is a randomized phase II open label study of daratumumab, weekly low-dose oral cyclophosphamide and dexamethasone with or without pomalidomide in patients with relapsed and refractory multiple myeloma. The study consists of two arms. Patients will be randomized into ARM A and ARM B in a 1:1 ratio.

In treatment ARM A patients will receive daratumumab, cyclophosphamide, dexamethasone and pomalidomide as per the following schedule:

* Daratumumab, IV, at 16 mg/kg, or Daratumumab, SC, at 1800 mg on days 1, 8, 15 and 22 for Cycles 1 and 2, on Days 1 and 15 for Cycles 3-6, and Day 1 of each cycle for Cycle 7 and beyond for each 28-day cycle.
* Cyclophosphamide, orally, at 400 mg on Days 1, 8, 15 of each 28-day cycle. In order to prevent myelotoxicity and bladder toxicity, cyclophosphamide will be discontinued after cycle 24.
* Dexamethasone orally at 20 mg on day of daratumumab administration (pre-daratumumab) and 20 mg on the following day. On weeks without daratumumab administration, 40 mg dexamethasone weekly.
* Pomalidomide, orally, at 4 mg on Days 1- 21 of each 28-day cycle.

In treatment ARM B, patients will receive daratumumab, cyclophosphamide, dexamethasone and pomalidomide as per the following schedule:

* Daratumumab, IV, at 16 mg/kg, or Daratumumab, SC, at 1800 mg on days 1, 8, 15 and 22 for Cycles 1 and 2, on Days 1 and 15 for Cycles 3-6, and Day 1 of each cycle for Cycle 7 and beyond for each 28-day cycle.
* Cyclophosphamide, orally, at 400 mg on Days 1, 8 and 15 of each 28-day cycle. In order to prevent myelotoxicity and bladder toxicity, cyclophosphamide will be discontinued after cycle 24.
* Dexamethasone at 20 mg orally on day of daratumumab administration (pre-daratumumab) and 20 mg on the following day. On weeks without daratumumab administration, 40mg dexamethasone weekly.
* Pomalidomide, orally, added at first progression at 4 mg on Days 1- 21 of each 28-day cycle.

Individual subjects will remain on treatment as long as there is no evidence of disease progression or unacceptable toxicity or patient/physician decision to discontinue. Disease assessment as determined by the Site Investigator will be made according to the IMWG response criteria guidelines for MM.

ELIGIBILITY:
Inclusion Criteria - Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Males or females, age 18 years or older.
2. ECOG performance status score of 0, 1 or 2.
3. Life expectancy of at least 3 months.
4. Measurable disease according to the IMWG criteria defined below. (These baseline laboratory studies for determining eligibility must be obtained during the screening period within 28 days prior to start of study drug):

   1. Serum monoclonal paraprotein (M-protein) ≥ 10 g/L (if IgG) or ≥5g/L (if IgA, D, E or M)
   2. Urine M-protein ≥ 200 mg/24 h
   3. Serum free light chains (FLC) assay: Involved FLC level ≥ 100 mg/L and an abnormal serum free light chain ratio (< 0.26 or > 1.65).
5. Relapsed or relapsed and refractory disease defined as documented disease progression during or after completing their last treatment line and it must have contained either a proteasome inhibitor and/or lenalidomide. The only exception for non-refractory patients is when re-treatment with these agents is medically contra-indicated.
6. Have undergone at least 1 prior line of therapy. Induction therapy followed by ASCT and consolidation/maintenance will be considered as one line.
7. Have achieved at least a Minimal Response (MR) or better to at least one previous line of therapy, as per IMWG response criteria.
8. Have received at least 2 consecutive cycles of prior treatment that have included lenalidomide or a proteasome inhibitor, either alone or in combination regimens, unless intolerant to these agents.
9. Subjects must be eligible for pomalidomide reimbursement by their provincial jurisdictions or by the criteria of their insurance companies.
10. The following laboratory results must be met within 10 days of first study drug adminitration:

    1. ANC ≥ 1.0 x 109/L
    2. Hemoglobin ≥ 80 g/L
    3. Platelets ≥ 70 x 109/L (or ≥50 x 109/L if ≥50% plasmacytosis in bone marrow.
    4. Calculated or measured CrCl ≥ 30 mL/min
    5. AST and ALT ≤ 3.0 x ULN
    6. Total bilirubin ≤ 2 x ULN unless known to have Gilbert's disease
    7. Corrected serum calcium ≤ 3.5 mmol/L
11. Have signed the informed consent documents indicating that the subject understands the purpose of and procedures required for the study and is willing to participate and adhere to the study protocol.
12. Females with child-bearing potential (FCBP†) must agree to use 2 reliable forms of contraception* simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including during dose interruptions), and for at least 90 days after study treatment discontinuation.

    †Females of childbearing potential (FCBP): a female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months).

    * The two methods of birth control used may be selected from the following categories, but the two methods cannot be selected from any one category: barrier method: i.e., condom (male or female) or diaphragm with spermicide; hormonal: i.e., contraceptive pill, patch; intrauterine device (IUD); vasectomy; or tubal ligation.
13. Females must agree to abstain from breastfeeding during study participation and 90 days after study drug discontinuation.
14. Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 90 days following discontinuation from this study, even if he has undergone a successful vasectomy.
15. Males must also agree to refrain from donating semen or sperm during the treatment phase and for 90 days after discontinuation from this study treatment.
16. All subjects must agree to refrain from donating blood while on study therapy and for 28 days after discontinuation from this study treatment.
17. All subjects must be eligible for enrollment and enrolled in the RevAid® program (refer to https://www.revaid.ca/revaid/ for RevAid eligibility).

Exclusion Criteria - Subjects who meet any of the following exclusion criteria are not eligible for enrollment:

1. Prior exposure to daratumumab (or other anti-CD38 monoclonal antibody) or pomalidomide.
2. History of prior allogeneic stem cell transplantation and showing evidence of active graft-versus-host disease or graft-versus-host disease that requires immunosuppressive therapy.
3. Chemotherapy or other anti-myeloma therapy within 14 days prior to the first dose of study drug.
4. Treatment-related toxicity that has not recovered ≤Grade 1 unless deemed to be irreversible (an example of an irreversible toxicity would include steroid induced cataracts). Peripheral neuropathy > Grade 2 or Grade 2 with pain will be excluded.
5. Subjects who have received steroids within 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy. Concomitant therapy medications that include corticosteroids are allowed if subject receive ≤ 10 mg of prednisone per day, or equivalent, as indicated for other medical conditions, or up to 100 mg of hydrocortisone as pre-medication for administration of certain medications or blood products prior to enrollment in this study.
6. Subjects who have received any investigational agents within 28 days or 5 half-lives (whichever is shorter, however the minimum allowed timeframe is 14 days) of the first dose (Cycle 1, Day 1).
7. Prior history of malignancies, other than MM, unless the subject has been free of the disease for 3 years or longer. Exceptions include the following:

   1. Basal or squamous cell carcinoma of the skin,
   2. Carcinoma in situ of the cervix or breast,
   3. Adenocarcinoma of the prostate (TNM stage of T1a or T1b).
8. Other concurrent severe and/or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection, acute diffuse pulmonary disease, pericardial disease, uncontrolled thyroid dysfunction) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol.
9. Known chronic obstructive pulmonary disease (COPD), defined as a FEV1 <50% predicted.
10. Known moderate or severe persistent asthma within the last 2 years, or currently has uncontrolled asthma of any classification.
11. History of or current uncontrolled cardiovascular disease including:

    1. Unstable angina, myocardial infarction, or known congestive heart failure Class III/IV (Appendix 5) within the preceding 12 months.
    2. Transient ischemic attack within the preceding 3 months, pulmonary embolism within the preceding 2 months.
    3. Any of the following: sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, cardiac arrest, Mobitz II second degree heart block or third degree heart block; known presence of dilated, hypertrophic, or restrictive cardiomyopathy.
    4. QTc prolongation as confirmed by ECG assessment at screening (QTc >470 milliseconds).
12. Women who are pregnant, breastfeeding or planning to become pregnant while enrolled in this study, or within 90 days after the last dose of study medications. Male subject who plans to father a child while enrolled in this study, within 90 days after the last dose of study medications.
13. Subjects who are:

    1. Known to be seropositive for human immunodeficiency virus (HIV).
    2. Seropositive for hepatits B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    3. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
14. Known allergies, hypersensitivity to mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the Daratumumab PM), or known sensitivity to mammalian-derived products.
15. Known CNS involvement, amyloidosis, or currently active plasma cell leukemia.
16. Subjects who are receiving any other investigational agent.
17. Autologous, peripheral stem cell transplant within 12 weeks of the first dose of study drug
18. Any other condition that, in the Investigator's opinion, would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 36 months of from randomization
  Progression-free survival evaluation after 36 months

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (11):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - CrossCancer Institute, Edmonton, Alberta
  - Fraser Valley Cancer Centre, Surrey, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre (Hamilton Health Sciences Centre), Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No